CLINICAL TRIAL: NCT00250640
Title: Open-label, Uncontrolled, Prospective Long-term Observation of Ventavis Inhalation Therapy in the Treatment of Patients With Primary Pulmonary Hypertension up to 4 Years
Brief Title: Observation of Patients With Primary Pulmonary Hypertension Receiving Prescribed Ventavis Inhalation Therapy Regarding Safety and Efficacy for up to 4 Years
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 91430; 308120 (Other: Company internal)
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Hypertension, Pulmonary
Keywords: Primary Pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Iloprost (Ventavis, BAYQ6256)

INTERVENTIONS:
Drug: Iloprost (Ventavis, BAYQ6256) — The recommended dose is 2.5 micrograms or 5.0 micrograms of inhaled iloprost (as delivered at the mouthpiece of the nebuliser). Dosing should follow the recommendations of the current package leaflet

SUMMARY:
This is an observational study to monitor the continued effectiveness of Ventavis (inhaled iloprost) in the long-term. The study observes the effects and the safety of Ventavis inhalation therapy over at least 2 years and up to 4 years. A total of 54 patients from around 30 study sites in Europe will be included in the study. This observational study will collect information in patients receiving a medication that is already available on prescription in the participating countries. Ventavis is used to treat moderate cases of primary pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* The treating physician has chosen Ventavis as a suitable long-term treatment for the patient
* Patient with primary pulmonary hypertension (i.e. Idiopathic Pulmonary Arterial Hypertension or Familial Pulmonary Arterial Hypertension) and classified as NYHA functional class III (NYHA = New York Heart Association)
* No prior treatment with Ventavis or other active treatments for primary pulmonary hypertension within 6 weeks of date of study inclusion (unless otherwise advised by Bayer Schering Pharma)

Exclusion Criteria:

* Any condition that prevents participation in the study, including pregnancy and other contraindications for Ventavis treatment (as listed in the current Ventavis Summary of Product Characteristics and patient package insert)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the disease in scope and the prescription of Ventavis mainly from expert clinics in the participating countries
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2005-04; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is 6-minute walking distance. Focus will lay on the individual changes (in meters) at Month 3 (after inhalation) compared to the value measured at baseline. | Month 3 Visit

SECONDARY OUTCOMES:
Relative change in the 6-minutes walking distance (%), as compared to baseline (BL): clinical improvement is defined as an increase of at least 10% vs BL; clinically significant deterioration is defined as a decrease of at least 30% vs BL. | all scheduled visits (Study period is min. 2 years and max. 4 years)
Changes in the NYHA class (to determine the patients' clinical conditions) vs. baseline will be classified into: improved, unchanged and deteriorated. Improvement is a negative difference; deterioration is a NYHA class increase from baseline. | all scheduled visits (Study period is min. 2 years and max. 4 years)
Mortality, defined as all-cause mortality, will be assessed for all patients included in this study. | all scheduled visits (Study period is min. 2 years and max. 4 years)
The safety and tolerability of Ventavis will be assessed by an examination of the adverse event data collected in this study. | all scheduled visits (Study period is min. 2 years and max. 4 years)
Other safety variable | At all scheduled visits (Study period is min. 2 years and max. 4 years)
  Weight, vital signs, findings in PPH-related signs and symptoms, hospitalization because of PPH, incidence of heart and/or lung transplantation
Other safety variables (optional assessment) | At all scheduled visits (Study period is min. 2 years and max. 4 years)
  Chest x-ray, electrocardiogram, findings of heart catheter test, findings of pulmonary function tests, findings of blood gas analyses

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (40):
- France (8):
  - Brest
  - Clamart
  - Lille
  - Lyon
  - Pessac
  - Reims
  - Strasbourg
  - Vandœuvre-lès-Nancy
- Germany (18):
  - Donaueschingen, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Löwenstein, Baden-Wurttemberg
  - Erlangen, Bavaria
  - München, Bavaria
  - Regensburg, Bavaria
  - Hamburg, Hamburg
  - Giessen, Hesse
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Homburg/Saar, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
  - Berlin, State of Berlin
  - Erfurt, Thuringia
- Italy (4):
  - Bologna
  - Pavia
  - Pisa
  - Roma
- Portugal (2):
  - Coimbra, Coimbra District
  - Lisbon
- Spain (4):
  - Barcelona, Barcelona
  - Córdoba, Córdoba
  - Barcelona
  - Madrid
- United Kingdom (4):
  - Glasgow
  - London
  - Newcastle upon Tyne
  - Sheffield